CLINICAL TRIAL: NCT00468221
Title: The Effect of Low Level Ozone Exposure on Healthy Volunteers
Acronym: Lowoz
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Environmental Protection Agency (EPA) (U.S. Federal Agency); National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Bradford Harris, MD, UNC_Chapel Hill
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 07-0304; R01ES012706 (NIH); R82952201
Record Dates: First submitted 2007-04-30; First posted 2007-05-02 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Healthy
Keywords: Ozone; Healthy Adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ozone Exposure — Low dose ozone exposure in chamber

SUMMARY:
The purpose of this research study is to learn more about the effects of 0.12 ppm ozone exposure on humans. We know from other studies that exposure to levels of ozone that are seen on bad air pollution days, can cause an increased risk of illness and even death in some people with certain health problems like asthma and heart disease. We also know from studies we have done in our lab that even healthy people can have an inflammatory (an increase in the amount of bacteria fighting cells) response to high levels of ozone. We suspect that exposure to low levels of ozone makes the body more susceptible to things like allergens. For instance, in persons allergic to pollen, exposure to ozone in the environment may cause them to have more allergy symptoms when they are around pollen than they would have if they were not exposed to ozone first. In this study we are looking to find the lowest level of ozone to which healthy people can be exposed without seeing that increased immune response. We will use 0.12 ppm ozone; this is roughly the amount of ozone you would be exposed to on a "yellow" ozone day in the triangle area in the summer if you spent the entire day out of doors and exercising moderately.

DETAILED DESCRIPTION:
Low levels of both endotoxin and O3 have been reported to prime airway responses for other stimuli, with a notable example being the immediate and late phase response to allergen. Likewise, epidemiological studies indicate that levels of O3 below the current air quality standards for ozone are still linked with exacerbation of respiratory tract disease. On a cellular level, both endotoxin and oxidants can prime inflammatory cells such that response to subsequently inhaled stimuli is enhanced. This has led to the idea that ozone may also enhance response to endotoxin and the reverse. As shown in our preliminary data, we have carefully examined the response to low levels of inhaled endotoxin and have found that a dose of 10,000 EU enhances the phagocytic function of macrophages, monocytes and PMNs and modifies the expression of cell surface receptors (CD11b, CD14), and alters IL-13 levels in sputum without causing PMN influx to the airway. This study is similar in design, but will evaluate the effects of ozone at a lower exposure level instead of endotoxin.

It has been thought that monocytes and macrophages did not mediate response to ozone because macrophages recovered from the airways of persons exposed to ozone had blunted responses to stimuli such as opsonized zymosan or other ligands, and in vitro, exposure of macrophages to ozone likewise renders them hypo-responsive to other stimuli, including endotoxin. There is general agreement that the airway response to endotoxin is mediated primarily by actions on macrophages and monocytes. However, monocytes undergo adaptation to endotoxin with previous challenge with endotoxin, and the chronic presence of endotoxin (i.e. in sepsis) also induces tolerance to the effect of additional exposure to endotoxin. Thus, suppression of monocyte/macrophage function by ozone may not be adequate evidence that these cells do not participate in ozone-induced airway inflammation.

It has also been argued that because ozone causes epithelial cells to generate mediators like IL-8 which is a potent chemoattractant for PMNs, the response to ozone was primarily orchestrated through these cells. However, there are data supporting a role for macrophages in response to ozone. Also, epithelial cells produce stress-induced endogenous ligands, many of which are known to be generated following exposure to ozone, which could interact with innate immune (e.g.CD14, TLR4), complement (e.g. CR3) or other receptors on airway mononuclear cells. An initial experiment by our group shows that ozone challenge of primary epithelial cell cultures (developed from nasal epithelial samplings of volunteers) yield supernatants which activate COX2 and induce IL-6 secretion from peripheral blood monocytes, indicating the potential for an O3-induced, epithelial-derived monocyte ligand. To approach the question of whether low level exposure to ozone modifies airway phagocyte biology (as determined primarily by cell surface marker expression, phagocyte function and endotoxin responsiveness), this study will be similar to the one detailed for endotoxin only volunteers are asked to undergo low level ozone exposure to determine if a priming dose can be identified that modifies monocyte biology but that is sub-threshold for inducing a neutrophil response in the airways.

Exposure to ozone as low as 0.12 ppm for 1 hour without exercise may prime response to allergen, yet is not an otherwise very effective dose for induction of inflammatory or lung function changes. 0.12 ppm O3 for 2 hours with 1 hour of intermittent exercise also does not yield airways inflammation but does result in generation of a salicylate product in volunteers dosed with aspirin which has been proposed as a marker of O3 exposure. Using these and similar studies as a guide, we will perform a study in which volunteers will undergo 0.12 ppm ozone exposure for 2 hours with moderate, intermittent exercise (to yield 35L/min ventilation for a total exercise duration of 1hr). We will examine sputum neutrophil levels (% PMNs and PMN/mg sputum), cell surface marker expression (CD11b, CD14) on sputum and blood inflammatory cells (monocytes, macrophages (sputum), phagocytosis and cytokine response to endotoxin stimulation, 6hr following exposure to ozone.

We will carry out an interim analysis after we have completed study in 6 volunteers to determine if we have identified a level of ozone that is likely to modify mononuclear cell function without significant neutrophilia. If 0.12 ppm of ozone for 2 hours appears to induce a priming response, no change in the PMN response and some modification of monocyte biology, we will continue with that dose. If we see an increase in PMNs, then we will refocus the protocol to challenge volunteers with 0.08 ppm O3 for 2 hours with moderate exercise. If there is no response at the macrophage level, then we would challenge volunteers with 0.2 ppm for 2 hours.

Multiple studies have linked ozone with increased morbidity and mortality. One possible explanation is decreased heart rate variability (HRV). In hospitalized patients, decreased HRV has been directly correlated with increased mortality under multiple conditions. Recent studies completed here have linked particulate matter to decreased HRV. In this study we will evaluate each subject's heart rate variability using ambulatory ECG monitoring.

Hypotheses

1. Low level ozone will prime airway macrophages/monocytes such that they will be more responsive to inflammatory stimuli, including endotoxin and opsonized zymosan.
2. Low level ozone will enhance airway and blood monocyte and macrophage function, and induce some alterations in some cell surface markers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Adult
* Nonsmoker
* Able to perform light exercise

Exclusion Criteria:

* Asthma
* active allergies
* chronic disease

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-06; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Inflammatory markers in sputum | post exposure

CONTACTS AND LOCATIONS:
Overall Officials: Bradford Harris, MD, Principal Investigator — University of North Carolina